CLINICAL TRIAL: NCT00627159
Title: ICA-CHAMP: Indo-Central Asian Cardiovascular Health Assessment and Management Program
Acronym: ICA-CHAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Charlotte Jones, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NRA3840015
Record Dates: First submitted 2008-01-14; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Cardiovascular Diseases; Hypertension; Hyperlipidemia
Keywords: community-based; culturally-sensitive; high risk assessment; education classes; cardiovascular risk profile; Indo-Asian population
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): high risk
  Interventions: Other: High risk assessment
- 2 (Other): low to moderate risk
  Interventions: Other: Low to moderate risk

INTERVENTIONS:
Other: High risk assessment — For all participants screened in the program, a cardiovascular risk profile is determined using information from the cardiovascular health history, blood pressure and cholesterol measurements, and The British Joint Societies Risk Prediction chart. All participants predicted to be at high risk are referred for assessment to a High Risk clinic in the community via the family doctor.
  Arms: 1
Other: Low to moderate risk — For all participants screened in the program, a cardiovascular risk profile is determined using information from the cardiovascular health history, blood pressure and cholesterol measurements, and The British Joint Societies Risk Prediction chart. All low to -moderate risk participants are directed to self-refer to the Calgary Health Region Multicultural education classes.
  Arms: 2

SUMMARY:
Research has shown that the presence of heart disease and stroke is higher in the Indo-Asian population compared to other ethno-cultural groups. This may be due to multiple reasons such as a higher presence of diabetes, high blood pressure, high cholesterol, obesity, and lower levels of physical activity.

This program will bring together the Calgary Indo-Central-Asian communities and the Calgary Healthcare community to help reduce the rate of heart disease and stroke through a supportive, culturally-sensitive program that is community-based through the following steps:

1. Increase awareness of heart disease and stroke through education among the Calgary Indo-Central-Asian population.
2. Identify early, the risk factors related to heart disease and stroke through screening programs.
3. Provide appropriate follow-up care to the population at risk for heart disease and stroke.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a leading cause of morbidity and mortality worldwide. Various studies have confirmed that individuals of SE Asian descent have a higher prevalence of cardiovascular disease compared with other ethnicities due to higher prevalence of metabolic syndrome, diabetes, insulin resistance, central obesity, dyslipidemias (lower high-density lipoprotein, increased lipoprotein[a], higher triglyceride levels), increased thrombotic tendency (increased plasminogen activator inhibitor-1 and decreased tissue plasminogen activator levels), and decreased levels of physical activity

Hypertension, in particular has become one of the leading causes of mortality among Asians. Projected figures suggest that in Indo-Asians hypertension prevalence will increase from 16.3% to 19.5% between 1995 and 2025. Despite increased prevalence of hypertension among Indo-Asians, the majority of cases remain undetected and poorly managed.

Disparities in health system utilization are associated with a high prevalence of hypertension leading to increased numbers of patients presenting with target organ damage such as stroke, heart failure and renal insufficiency. Epidemiological studies have demonstrated that high-risk ethnic groups have access barriers to mainstream programs and may benefit from targeted and culture specific interventions. Given that Indo-Asians represent an increasing proportion of the Canadian population and are at higher risk of cardiovascular diseases and experience health care access barriers, the initiation of an tailored risk factor screening and intervention program is timely.

The collaborative effort between the target communities and the healthcare system provides an unique opportunity to develop and evaluate a sustainable screening, early detection and intervention program in hypertension and other CVD risk factors, tailored to meet the unique cultural needs of the target population. Only an all encompassing program of this scope will reduce the risk of cardiovascular diseases in this highly susceptible population.

The project objectives are as follows:

* To increase Indo-Central Asian community awareness of cardiovascular risk factors
* To develop and implement a community based, culturally sensitive and self-sustaining cardiovascular risk factor screening and management program.
* To increase early detection of modifiable, undiagnosed, and uncontrolled cardiovascular risk factors
* Using a partnership-based, culturally appropriate and integrated approach, provide a sustainable and cost effective intervention program for optimal management of risk factors in the Indo-Central Asian population utilizing existing health region and community resources.
* To develop a continuum of care that addresses the needs of Indo-Central Asian Calgarians and that tailors the intensity of intervention to the perceived risk
* To validate the "Continuum of Care" process

The project components are as follows:

* Screening sessions: The project will utilize a previously developed Indo-Asian Diabetes Initiative methodology to recruit and train volunteers from the target community. Using standardized interview questions, the following information will be collected: age, gender, family history (first degree relative with premature cardiovascular disease), and other cardiovascular risk factors. Trained volunteers would administer the questions during one to one interviews in English or a common language used by the participant in the community. Blood pressures will be obtained using a validated Bp assessment tool (BpTRU). All those screened that have either high blood pressure (≥140/90 or ≥130/80 with diabetes) or at least one risk factor (positive family or personal history of cardiovascular disease, diabetes, smoker, known elevated cholesterol or on medications for HBP, lipids or diabetes) will then go on to have capillary measurements of random TC/HDL performed by the Cholestech desktop reflometer (Hayward CA).

Based on health history and assessments obtained, the total CVD risk (coronary heart disease and stroke) will be predicted using the Joint British Societies Cardiovascular Disease Risk Prediction Chart. Those participants found to be high risk (>20 % 10 year CVD risk) will be referred, via the family physician, to a HRIC clinic. Those at moderate or low risk (≤20% 10 year CVD risk) will be referred to the CDM program. All participants that are screened will receive the adapted and culturally sensitive versions of the 2007 Canadian Public Recommendations education booklet (adapted by Blood Pressure Canada) that includes hypertension, dietary, alcohol and smoking cessation information.

* Intervention: All qualifying participants will be assessed by a volunteer pharmacist, nurse, physician, or other health care professional who will review the participants' current medications and provide education around adherence and adverse events. The completed assessments and the predicted risk scores will be reviewed with the participant. The predicted risk score will facilitate the participant's enrolment in the appropriate follow up program. Participants will be re-directed back to the family physician for BP monitoring and medication initiation or adjustment as required. Participants will be provided with a "Health Report" that will include their current medications, blood pressures, TC and HDL results, predicted CVD risk score and follow-up instructions. Interventions will be as follows:

  * High CVD Risk Intervention: Individuals at high risk will be referred to a High Risk Intervention Clinic for full cardiovascular evaluation. This includes a history and physician exam by an Internal Medicine Specialist or alternate specialist with similar cardiovascular training and experience An ECG will be performed and likely either a stress test or nuclear cardiology study. Risk factors will be aggressively managed.
  * Low and Moderate CVD Risk Intervention: Individuals at low or moderate risk will be referred to a convenient and culturally appropriate CDM community program (culturally sensitive education and physical activity programs).
* Follow-up Sessions: Consenting participants will be contacted by a project volunteer and be invited back for reassessment one year after initial evaluation. Reassessment will entail a work-up similar to that conducted during the initial screening session.

ELIGIBILITY:
Inclusion Criteria:

* Indo-Cental Asian decent
* Minimum 45 years of age
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Current cardiology specialist

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Baseline and one year change in blood pressure and total cholesterol, HDL cholesterol and TC/HDL ratio (High and low to moderate risk program participants) | one year

SECONDARY OUTCOMES:
Cardiovascular risk profile and risk scores (Joint British Societies Cardiovascular Disease Risk Prediction Chart) of all participants at baseline and upon completion of the High Risk Assessment and Calgary Health Region Multicultural education programs. | one year
Baseline profiles of attendees versus no-shows at both High Risk Assessment clinics and Calgary Health Region Multicultural education programs | one year
"No-show" rates at High Risk Assessment clinics and Calgary Health Region Multicultural education program vs. historical rates. | one year
Proportion of High Risk Assessment Clinic attendees identified as having occult Coronary Artery Disease and requiring angioplasty and/or Coronary Artery Bypass Graft. | one year
Post Hoc variation of the Joint British Societies Cardiovascular Disease Risk Prediction Chart versus ETHRISK | one year
Participant and community leader/volunteer satisfaction with the program | one year
Participant opinion regarding usefulness of the culturally-sensitive educational information provided at the screening session. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte - Jones, PhD, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Hindu Society of Calgary, Calgary, Alberta
  - Dashmesh Cultural Centre, Calgary, Alberta

REFERENCES:
- [Background] Bedi US, Singh S, Syed A, Aryafar H, Arora R. Coronary artery disease in South Asians: an emerging risk group. Cardiol Rev. 2006 Mar-Apr;14(2):74-80. doi: 10.1097/01.crd.0000182411.88146.72. PMID 16493244
- [Background] Aarabi M, Jackson PR. Predicting coronary risk in UK South Asians: an adjustment method for Framingham-based tools. Eur J Cardiovasc Prev Rehabil. 2005 Feb;12(1):46-51. PMID 15703505
- [Background] Anand SS, Yusuf S, Vuksan V, Devanesen S, Teo KK, Montague PA, Kelemen L, Yi C, Lonn E, Gerstein H, Hegele RA, McQueen M. Differences in risk factors, atherosclerosis, and cardiovascular disease between ethnic groups in Canada: the Study of Health Assessment and Risk in Ethnic groups (SHARE). Lancet. 2000 Jul 22;356(9226):279-84. doi: 10.1016/s0140-6736(00)02502-2. PMID 11071182
- [Background] Davachi S, Flynn M, Edwards A. A health region/community partnership for Type 2 diabetes risk factor screening in Indo-Asian communities. Canadian Journal of Diabetes 29(2):87-94, 2005.
- [Background] Brindle P, May M, Gill P, Cappuccio F, D'Agostino R Sr, Fischbacher C, Ebrahim S. Primary prevention of cardiovascular disease: a web-based risk score for seven British black and minority ethnic groups. Heart. 2006 Nov;92(11):1595-602. doi: 10.1136/hrt.2006.092346. Epub 2006 Jun 8. PMID 16762981
- [Background] British Cardiac Society; British Hypertension Society; Diabetes UK; HEART UK; Primary Care Cardiovascular Society; Stroke Association. JBS 2: Joint British Societies' guidelines on prevention of cardiovascular disease in clinical practice. Heart. 2005 Dec;91 Suppl 5(Suppl 5):v1-52. doi: 10.1136/hrt.2005.079988. No abstract available. PMID 16365341
- See also: Related Info — http://www.hypertension.ca
- See also: Related Info — http://www.heartandstroke.ca